CLINICAL TRIAL: NCT07298668
Title: Standard Modifiable Risk Factors in Middle Eastern Patients With Stroke (Jo-SMMART Study)
Brief Title: Cardiovascular Risk Factors in Middle Eastern Patients With Stroke
Acronym: JoSMMART
Status: Not yet recruiting | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: JOCVA1.NOV2025/2
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Low-Density-Lipoprotein-cholesterol Level; Risk Factors
Keywords: Stroke; Risk factors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is a well-known a leading cause of death and disability in the Middle East. There remain many knowledge gaps in evaluating the prevalence of risk factors among patients with stroke in the Middle East. Unravelling the impact of these risk factors and controlling them can positively lower the incidence of stroke. Disparities in stroke risk factors, may well be related to ethnicity of the Middle Eastern populations , will be compared with those among stroke patients in the western literature.

DETAILED DESCRIPTION:
Stroke is a well-known a leading cause of death and disability in the Middle East. There remain many knowledge gaps in evaluating the prevalence of risk factors among patients with stroke in the Middle East. Unravelling the impact of these risk factors and controlling them can positively lower the incidence of stroke. Disparities in stroke risk factors, may well be related to ethnicity of the Middle Eastern populations , will be compared with those among stroke patients in the western literature.

These clinically relevant issues have not been studied extensively in the Middle East where most of the studies in atherosclerotic cardiovascular disease have focused on acute coronary syndrome more than stroke. Exploring new information on risk factors of stroke in this region that helps fill some of the knowledge gaps.

Stroke has been attributed, in the majority of cases, to the traditional four standard modifiable risk factors of hypertension, type 2 diabetes, dyslipidemia, and cigarette smoking. However, ethnicity and geography account for the interregional differences of the prevalence of risk factors in patients with stroke.

The Jo-SMMART ill evaluate risk factors in 2000 stroke patients in Jordan as a representative of the Middle Eastern population, the prevalence of those with none of the 4 risk factors and the differences in clinical profiles and demographic features on those with risk factors and those with no risk factors. Lipid profile and use of lipid lowering agents will also be evaluated, and furthermore the die0fferneces between young vs old, and men vs women stroke patients ill be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke upon admission to the hospital
* Adult aged 18 years or older
* Available lipid profile on hospital admission

Exclusion Criteria:

* Stroke diagnosis unconfirmed
* age younger than 18 years
* No available lipid profile on admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Will enroll adults admitted to the hospital with a working diagnosis of stroke and then the diagnosis is confirmed by a neurologist. Patients ii be interviewed for data collection of 4 risk factors as above in addition to the serum level of LDLC and the use of lipid lowering agents.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypertension in stroke patients (survey interview) | Baseline
  BP more 140/90 or known diagnosis of high blood pressure or patient already on blood pressure medication
Prevalence of type 2 diabetes in stroke patients (survey interview) | BASELINE
  HbA1c more than 6.5%, or known diagnosis of type 2 diabetes or patient already on anti diabetes medications
Prevalence of elevated serum level of low density lipoprotein cholesterol in stroke patients (survey interview) | BASELINE
  Elevated serum level of low density lipoprotein cholesterol > 55 mg/dl or patient already on lipid lowering medication
Prevalence of current cigarette smoking in stroke patients (survey interview) | BASELINE
  Known current cigarette smoking of any number of cigarettes per day
Use of lipid lowering therapy (survey interview) | BASELINE
  Current use of statin, ezitimibe, PCS9 inhibitor of small interfering RNA agent to lower the LDL-C

CONTACTS AND LOCATIONS:
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be available in the form of excel sheet with no disclosure of patients names. Can be requested from the study director